CLINICAL TRIAL: NCT02496767
Title: A Phase 3, Multi-National, Double-Blind, Randomized, Placebo-Controlled, Stratified, Parallel Group, Study to Evaluate the Safety, Tolerability and Efficacy of Tirasemtiv in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Ventilatory Investigation of Tirasemtiv and Assessment of Longitudinal Indices After Treatment for a Year
Acronym: VITALITY-ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CY 4031; 2014-005413-23 (EudraCT Number)
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: fast skeletal troponin activator; tirasemtiv; CK-2017357; double-blind; randomized; placebo-controlled
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - Placebo (Placebo Comparator): Day 1 through Week 48: 2 placebo tablets twice daily
  Interventions: Drug: Placebo tablets
- Group 2 - 250 mg tirasemtiv (Experimental): Day 1 through Week 48: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM
  Interventions: Drug: Tirasemtiv; Drug: Placebo tablets
- Group 3 - 375 mg tirasemtiv (Experimental): Day 1 through Week 2: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM; Weeks 3 through 48: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
  Interventions: Drug: Tirasemtiv; Drug: Placebo tablets
- Group 4 - 500 mg tirasemtiv (Experimental): Day 1 through Week 2: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in PM; Weeks 3 and 4: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM; Weeks 5 through 48: 2 tablets of tirasemtiv (250 mg) in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
  Interventions: Drug: Tirasemtiv; Drug: Placebo tablets

INTERVENTIONS:
Drug: Tirasemtiv
  Other Names: CK-2017357
  Arms: Group 2 - 250 mg tirasemtiv; Group 3 - 375 mg tirasemtiv; Group 4 - 500 mg tirasemtiv
Drug: Placebo tablets

SUMMARY:
This study assessed the effect of tirasemtiv versus placebo on respiratory function in patients with ALS.

DETAILED DESCRIPTION:
CY 4031 was a multi-national, double-blind, randomized, placebo-controlled, stratified, parallel group study of tirasemtiv in patients with ALS. The study had three phases: an open-label phase (2 weeks), a double-blind, placebo-controlled phase (48 weeks), and a double-blind, placebo-controlled tirasemtiv withdrawal phase (4 weeks). Patients who completed 2 weeks of treatment with open-label tirasemtiv (125 mg twice daily) were randomized 3:2:2:2 to placebo or one of three dose levels of tirasemtiv (250 mg/day, 375 mg/day, or 500 mg/day). Approximately 600 patients were planned to be enrolled into the open-label treatment phase.

Patients taking riluzole at study entry could continue use of riluzole during the study as long as they had been on a stable dose for at least 30 days prior to study screening. In addition, for patients randomized to tirasemtiv, the riluzole dose was reduced to half the approved dose (ie, reduced to 50 mg once daily) because administration of tirasemtiv approximately doubles the exposure to concomitant riluzole. Patients randomized to placebo continued riluzole at 50 mg twice daily. This was accomplished without unmasking the study's blind as follows:

1. All patients on riluzole took their morning 50 mg dose of riluzole from their personal riluzole supply.
2. The sponsor supplied the evening riluzole dose as double-blind study medication, as follows: (a) for patients randomized to placebo, the double-blind, evening riluzole dose was 50 mg of active riluzole; (b) for patients randomized to tirasemtiv, the double-blind, evening riluzole dose was a matching placebo for riluzole.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of familial or sporadic ALS (defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria) ≤ 24 months prior to screening
* Upright SVC ≥ 70 % of predicted for age, height and sex
* Able to swallow tablets without crushing, and in the opinion of the Investigator, is expected to continue to be able to do so during the trial
* A caregiver if one is needed
* Clinical laboratory findings within the normal range or, if outside the normal range, deemed not clinically significant by the Investigator
* Male patients must agree for the duration of the study and 10 weeks after the end of the study to use a condom during sexual intercourse with female partners who are of childbearing potential (i.e., following menarche until post-menopausal if not anatomically and physiologically incapable of becoming pregnant) and to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide, or oral contraceptives) or the male patient must agree to abstain from sexual intercourse during and for 10 weeks after the end of the study, unless the male patient has had a vasectomy and confirmed sperm count is zero
* Female patients must be post-menopausal (≥ 1 year) or sterilized, or, if of childbearing potential, not be breastfeeding, have a negative pregnancy test, have no intention to become pregnant during the course of the study, and use effective contraceptive drugs or devices while requiring male partner to use a condom for the duration of the study and for 10 weeks after the end of the study
* Patients must be either on a stable dose of riluzole 50 mg twice daily for at least 30 days prior to screening or have not taken riluzole for at least 30 days prior to screening and are willing not to begin riluzole use until they complete study drug dosing

Exclusion Criteria:

* At the time of screening, any use of non-invasive positive pressure ventilation (NIPPV, e.g. continuous positive airway pressure [CPAP] or bi-level positive airway pressure [BiPAP]) for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation
* Patients with a diaphragm pacing system (DPS) at study entry or who anticipate DPS placement during the course of the study
* BMI of 20.0 kg/m2 or lower
* Unwilling or unable to discontinue tizanidine and theophylline-containing medications during study participation
* Serum chloride outside the normal reference range
* Neurological impairment due to a condition other than ALS, including history of transient ischemic attack within the past year
* Presence at screening of any medically significant cardiac, pulmonary, GI, musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or efficacy data, including, but not limited to:

  1. Poorly controlled hypertension
  2. NYHA Class II or greater congestive heart failure
  3. Chronic obstructive pulmonary disease or asthma requiring daily use bronchodilator medications
  4. GI disorder that might impair absorption of study drug
  5. History of significant liver disease defined by bilirubin > 2 times the upper limit of normal (ULN) or ALT or AST > 3 times the ULN on repeat testing
  6. Poorly controlled diabetes mellitus
  7. History of vertigo within three months of study entry
  8. History of syncope without an explainable or treated cause
  9. History of untreated intracranial aneurysm or poorly controlled seizure disorder
  10. Amputation of a limb
  11. Cognitive impairment, related to ALS or otherwise, sufficient to impair the patient's ability to give informed consent and to understand and/or comply with study procedures
  12. Cancer with metastatic potential (other than basal cell carcinoma, carcinoma in situ of the cervix, or squamous cell carcinoma of the skin excised with clean margins) diagnosed and treated within the last two years
  13. Any other condition, impairment or social circumstance that, in the opinion of the Investigator, would render the patient not suitable to participate in the study
  14. Patient judged to be actively suicidal or a suicide risk by the Investigator
* Has taken any investigational study drug within 30 days or five half-lives of the prior agent, whichever is greater, prior to dosing
* Prior participation in any form of stem cell therapy for the treatment of ALS
* Previously received tirasemtiv in any previous clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Cytokinetics
Locations (81):
- United States (49):
  - St. Joseph's Hospital & Medical Center - Barrow Neurology Clinics, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Carol and Frank Morsini Center for Advanced Health Care - University of South Florida, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Hospital and Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Neurology Associates, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center Dept of Neurology, Lebanon, New Hampshire
  - Hospital for Special Surgery, New York, New York
  - Neurological Institute Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Neurosciences Institute: Neurology - Charlotte, Charlotte, North Carolina
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Brain and Spine Institute ALS Center, Portland, Oregon
  - Oregon Health and Science Center, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Penn Comprehensive Neuroscience Center, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Virgina Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University Department of Neurology, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital, Department of Neurology, Milwaukee, Wisconsin
- UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant, Belgium
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - Edmonton Kaye Clinic, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QE II Health Sciences Centre, NHI Site, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Notre-Dame Hospital/CHUM, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Quebec - Universite Laval Hopital de l'Enfant-Jesus, Québec
- France (7):
  - Hopital R. Salengro, CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Hopital de la Timone, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - CHU de Nice - Hopital Pasteur 2, Nice
  - Hopital de la Salpetriere, Paris
  - Bretonneau University Hospital, Tours
- Germany (3):
  - University of Ulm, Department of Neurology, Ulm, Baden-Wurttemberg
  - Hannover Medical School, Department of Neurology, Hanover, Lower Saxony
  - Charite Campus Virchow-Klinikum, Neurology Department, Berlin
- Clinical Research Centre, Beaumont Hospital, Dublin, Ireland
- Italy (3):
  - IRCCS Istituto Auxologico Italiano - U.O. Neurologia, Milan
  - Centro Clinico NEMO - Fondazione Serena Onlus, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Dipartimento di Neuroscienze "Rita Levi Moltalcini" A.O.U. Citta della Salute e della Scienza di Torino P.O. "Molinette", Torino
- University Medical Center Utrecht, Utrecht, Netherlands
- Hospital Santa Maria-Centro Hospitalar Lisboa Norte, Lisbon, Portugal
- Hospital San Rafael, Madrid, Spain
- United Kingdom (4):
  - Derriford Hospital, Plymouth, Devon
  - Walton Centre for Neurology and Neurosurgery, Liverpool
  - Clinical Research Centre, Royal London Hospital, London
  - Kings College Hospital, London

REFERENCES:
- [Derived] Simkins TJ, Kupfer S, Malik FI, Meng L, Rudnicki SA, Wei J, Shefner JM, Bowser R. Plasma neurofilament analysis in VITALITY-ALS. Amyotroph Lateral Scler Frontotemporal Degener. 2025 Feb;26(1-2):103-112. doi: 10.1080/21678421.2024.2423707. Epub 2024 Nov 8. PMID 39513379
- [Derived] Andrews JA, Cudkowicz ME, Hardiman O, Meng L, Bian A, Lee J, Wolff AA, Malik FI, Shefner JM. VITALITY-ALS, a phase III trial of tirasemtiv, a selective fast skeletal muscle troponin activator, as a potential treatment for patients with amyotrophic lateral sclerosis: study design and baseline characteristics. Amyotroph Lateral Scler Frontotemporal Degener. 2018 May;19(3-4):259-266. doi: 10.1080/21678421.2018.1426770. Epub 2018 Feb 6. PMID 29402141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with familial or sporadic amyotrophic lateral sclerosis were enrolled at 79 sites in Belgium, Canada, France, Germany, Great Britain, Ireland, Italy, Netherlands, Portugal, Spain, and the United States. The first patient was screened on 03 September 2015 and the last subject completed on 27 September 2017.
Pre-assignment Details: All enrolled patients began open-label tirasemtiv (250 mg) in a 2-week lead-in phase. Completed patients were randomized (3:2:2:2) to placebo or tirasemtiv (250, 375, or 500 mg) for 48 weeks of double-blind treatment. After which, patients on tirasemtiv were re-randomized (1:1) to placebo or tirasemtiv (current dose) for a 4-week withdrawal phase.
Groups:
- Open-label Lead-in: 250 mg Tirasemtiv: Open-label tirasemiv (125 mg twice daily) for 2 weeks
- Double-blind, Placebo-controlled: Group 1 - Placebo: Day 1 through Week 48: 2 placebo tablets twice daily
- Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv: Day 1 through Week 48: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM
- Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv: Day 1 through Week 2: 1 tablet (125 mg) of tirasemtiv and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM; Weeks 3 through 48: 1 tablet (125 mg) of tirasemtiv and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
- Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv: Day 1 through Week 2: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM; Weeks 3 and 4: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM; Weeks 5 through 48: 2 tablets of tirasemtiv (250 mg) in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
- Double-blind, Withdrawal: Placebo: Following the 48-week double-blind, placebo-controlled phase of the study, patients in the placebo group continued placebo for an additional 4 weeks.
- Double-blind, Withdrawal: Tirasemtiv to Placebo: Following the 48-week double-blind, placebo-controlled phase of the study, approximately half the patients in a tirasemtiv group were re-randomized to placebo treatment for 4 weeks.
- Double-blind, Withdrawal: Tirasemtiv: Following the 48-week double-blind, placebo-controlled phase of the study, approximately half the patients in a tirasemtiv group were re-randomized to remain on tirasemtiv treatment (at the same dose received at the end of the double-blind, placebo-controlled phase) for 4 weeks.
Period: Open-label Lead-in Phase
Arm/Group | Open-label Lead-in: 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv | Double-blind, Withdrawal: Placebo | Double-blind, Withdrawal: Tirasemtiv to Placebo | Double-blind, Withdrawal: Tirasemtiv
Started | 744 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 565 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 179 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 176 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind, Placebo-controlled Phase
Arm/Group | Open-label Lead-in: 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv | Double-blind, Withdrawal: Placebo | Double-blind, Withdrawal: Tirasemtiv to Placebo | Double-blind, Withdrawal: Tirasemtiv
Started | 0 | 188 | 126 | 126 | 125 | 0 | 0 | 0
Completed | 0 | 132 | 80 | 65 | 59 | 0 | 0 | 0
Not Completed | 0 | 56 | 46 | 61 | 66 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 13 | 23 | 43 | 43 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 13 | 9 | 8 | 14 | 0 | 0 | 0
Not completed — Death | 0 | 10 | 6 | 2 | 4 | 0 | 0 | 0
Not completed — Various | 0 | 9 | 4 | 5 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 3 | 1 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind, Withdrawal Phase
Arm/Group | Open-label Lead-in: 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv | Double-blind, Withdrawal: Placebo | Double-blind, Withdrawal: Tirasemtiv to Placebo | Double-blind, Withdrawal: Tirasemtiv
Started | 0 | 0 | 0 | 0 | 0 | 132 | 103 | 101
Completed | 0 | 0 | 0 | 0 | 0 | 126 | 99 | 96
Not Completed | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 5
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics are provided for the Full Analysis Set, comprised of patients who received at least 1 dose of study drug during the randomized double-blind, placebo-controlled phase and had at least 1 post-randomization efficacy assessment (totaling 561 patients: 188, 126, 125, and 122 patients in Groups 1, 2, 3, and 4, respectively).
Groups:
- Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv: Day 1 through Week 2: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM; Weeks 3 through 48: 1 tablet (125 mg) of tirasemtiv and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
- Total: Total of all reporting groups
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv | Total
Number analyzed (Participants) | 188 | 126 | 125 | 122 | 561
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.63) | 57.1 (10.20) | 57.4 (9.09) | 56.0 (10.81) | 56.5 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 30 | 42 | 38 | 175
  Male | 123 | 96 | 83 | 84 | 386
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 0 | 2 | 1 | 6
  White | 181 | 123 | 120 | 117 | 541
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Riluzole use at baseline [Count of Participants; unit: Participants] | 141 | 95 | 94 | 92 | 422

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 of the Double-blind, Placebo-controlled Phase in Percent Predicted Slow Vital Capacity (SVC)
Description: SVC was measured using a spirometer (in units of liters). Following 3 to 5 breaths at rest, the patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs). Values obtained were converted to % predicted values (ie, the test result as a percent of predicted values for patients of similar demographic and baseline characteristics [eg, height, age, sex], based on Knudson 83 normative values).
Time Frame: 24 weeks
Population: The data presented are for the Full Analysis Set, comprised of patients who received at least 1 dose of study drug during the randomized double-blind, placebo-controlled phase and had at least 1 post-randomization efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: % predicted
Groups:
- Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv: Day 1 through Week 2: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the PM; Weeks 3 through 48: 1 tablet of tirasemtiv (125 mg) and 1 tablet of matching placebo in the AM and 2 tablets of tirasemtiv (250 mg) in the PM
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
% predicted | -14.354 (1.2270) | -12.648 (1.5165) | -13.742 (1.6076) | -13.927 (1.7213)
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.3782, Repeated-measures mixed model; Least squares mean difference = 1.707, 95% CI 2-sided [-2.089 to 5.503], Standard Error of Mean 1.9365
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.7625, Repeated-measures mixed model; Least squares mean difference = 0.612, 95% CI 2-sided [-3.359 to 4.583], Standard Error of Mean 2.0245
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.8394, Repeated-measures mixed model; Least squares mean difference = 0.428, 95% CI 2-sided [-3.711 to 4.566], Standard Error of Mean 2.1081

2. Secondary Outcome: Change From Baseline in the ALSFRS-R Respiratory Domain Score at the End of 48 Weeks of Double-blind, Placebo-controlled Treatment
Description: The ALSFRS-R is used to measure the progression and severity of disease; it consists of 12 questions, assessing a patient's capability and independence in functional activities relevant to ALS, categorized in 4 domains: bulbar functions, fine motor tasks, gross motor tasks, and respiratory function. Respiratory function consists of 3 of the 12 questions, which assess dyspnea, orthopnea, and respiratory insufficiency. Each question is scored from 0 (indicating incapable or dependent) to 4 (normal). The sum of the response to these 3 questions represents the respiratory domain score. The respiratory domain score ranges from 0 to 12, with higher scores reflecting more normal function and lower scores reflecting more impaired function.
Time Frame: 48 weeks
Population: The data provided are for the Full Analysis Set, comprised of patients who received at least 1 dose of study drug during the randomized double-blind, placebo-controlled phase and had at least 1 post-randomization efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
units on a scale | -2.26 (0.258) | -1.95 (0.320) | -2.41 (0.340) | -2.59 (0.355)
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.4521, Repeated-measures mixed model; Least squares mean difference = 0.31, 95% CI 2-sided [-0.50 to 1.12], Standard Error of Mean 0.410
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.7120, Repeated-measures mixed model; Least squares mean difference = -0.16, 95% CI 2-sided [-1.00 to 0.68], Standard Error of Mean 0.426
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.4510, Repeated-measures mixed model; Least squares mean difference = -0.33, 95% CI 2-sided [-1.19 to 0.53], Standard Error of Mean 0.439

3. Secondary Outcome: Slope of Mega-score of Muscle Strength During the 48 Weeks of Double-blind, Placebo-controlled Treatment
Description: A hand-held dynomometer, with a scale of 0 to 300 pounds, was used to measure muscle strength and handgrip strength (bilateral); the muscle groups tested were: elbow flexion (bilateral), wrist extension (bilateral), knee extension (bilateral), and ankle dorsiflexion (bilateral). The muscle strength mega-score was calculated as the average of responses to all tested muscles as well as handgrip strength. The slope of muscle strength mega-score was the change over time (48 weeks) and analyzed using a mixed model that assumed a random slope effect. For this endpoint, negative values indicate a decline in muscle strength over time.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: pounds/day
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
pounds/day | -0.1501 [-0.1729 to -0.1272] | -0.1512 [-0.1794 to -0.1230] | -0.1434 [-0.1742 to -0.1126] | -0.1413 [-0.1730 to -0.1095]
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.9505, Repeated-measures mixed model; Mean Difference (Final Values) = -0.0011, 95% CI 2-sided [-0.0374 to 0.0351]
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.7336, Repeated-measures mixed model; Mean Difference (Final Values) = 0.0066, 95% CI 2-sided [-0.0317 to 0.0450]
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.6593, Repeated-measures mixed model; Mean Difference (Final Values) = 0.0088, 95% CI 2-sided [-0.0303 to 0.0479]

4. Secondary Outcome: Time to the First Occurrence of a Decline From Baseline in Percent Predicted SVC ≥ 20 Percentage Points or the Onset of Respiratory Insufficiency or Death All 48 Weeks of Double-blind, Placebo-controlled Treatment
Description: This endpoint evaluated the time to occurrence of a decline in percent predicted SVC (as measured by spirometry) of ≥ 20 percentage points, or the onset of respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥ 22 hours per day for ≥10 consecutive days), or death, whichever was first, during the 48-week double-blind, placebo-controlled treatment phase.
  Note: The median time to a ≥ 20% decline in percent predicted SVC, onset of respiratory insufficiency, or death was 302 days for the placebo group and 359, 334, and 337 days for the 250 mg, 375 mg, and 500 mg tirasemtiv groups, respectively. The data presented for this endpoint are the number and percent of patients who met the endpoint.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
Participants | 98 | 58 | 58 | 57
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.2369, Regression, Cox; Hazard Ratio (HR) = 0.818, 95% CI 2-sided [0.587 to 1.141] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.9420, Regression, Cox; Hazard Ratio (HR) = 0.988, 95% CI 2-sided [0.711 to 1.372] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.6853, Regression, Cox; Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.668 to 1.304] — Hazard ratio for tirasemtiv vs placebo

5. Secondary Outcome: Time to the First Occurrence of a Decline in SVC to ≤ 50% Predicted, or the Onset of Respiratory Insufficiency, or Death During the 48 Weeks of Double-blind, Placebo-controlled Treatment
Description: This endpoint evaluated the time to occurrence of a decline in SVC (as measured by spirometry) to ≤ 50% predicted, or the onset of respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥ 22 hours per day for ≥10 consecutive days), or death, whichever was first, during the 48-week double-blind, placebo-controlled treatment phase.
  Note: The median time to a decline in SVC to ≤ 50% predicted, onset of respiratory insufficiency, or death was not estimable for the placebo group or the 375 mg tirasemtiv group. The median time was estimated as 363 and 351 days for the 250 mg and 500 mg tirasemtiv groups, respectively. The data presented for this endpoint are the number and percent of patients who met the endpoint.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
Participants | 57 | 39 | 30 | 32
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.7667, Regression, Cox; Hazard Ratio (HR) = 1.066, 95% CI 2-sided [0.698 to 1.627] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.6619, Regression, Cox; Hazard Ratio (HR) = 0.904, 95% CI 2-sided [0.577 to 1.419] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.5856, Regression, Cox; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.561 to 1.386] — Hazard ratio for tirasemtiv vs placebo

6. Secondary Outcome: Change From Baseline in the ALSFRS-R Total Score to the End of 48 Weeks of the Double-blind, Placebo-controlled Treatment
Description: The ALSFRS-R is used to measure the progression and severity of disease; it consists of 12 questions, assessing a patient's capability and independence in functional activities relevant to ALS, categorized in 4 domains: gross motor tasks, fine motor tasks, bulbar functions, and respiratory function. Each question is scored from 0 (indicating incapable or dependent) to 4 (normal). The total score ranges from 0 to 48, with higher scores reflecting more normal function and lower scores reflecting more impaired function.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
units on a scale | -11.39 (0.695) | -11.39 (0.859) | -12.19 (0.903) | -11.99 (0.937)
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.9991, Repeated-measures mixed model; Least squares mean difference = 0.00, 95% CI 2-sided [-2.17 to 2.17], Standard Error of Mean 1.103
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.4808, Repeated-measures mixed model; Least squares mean difference = -0.80, 95% CI 2-sided [-3.04 to 1.43], Standard Error of Mean 1.138
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv; Test type: Superiority; p = 0.6082, Repeated-measures mixed model; Least squares mean difference = -0.60, 95% CI 2-sided [-2.89 to 1.69], Standard Error of Mean 1.165

7. Secondary Outcome: Time to the First Use of Mechanical Ventilatory Assistance or Death During All 48 Weeks of Double-blind, Placebo-controlled Treatment
Description: This endpoint evaluated the time to occurrence of mechanical ventilatory assistance (defined as invasive or non-invasive ventilation for at least 2 hours over a 24-hour period for at least 5 consecutive days) or death, whichever was first, during the 48-week double-blind, placebo-controlled treatment phase.
  Note: The median time to first use of mechanical ventilatory assistance or death was not estimable for all but the 375 mg tirasemtiv group (with a value of 367 days). As such the number and percent of patients who met the endpoint (ie, had mechanical ventilatory assistance or died) are presented.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv
Number analyzed (Participants) | 188 | 126 | 125 | 122
Participants | 60 | 31 | 37 | 33
Statistical Analysis 1: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv; Test type: Superiority; p = 0.2602, Regression, Cox; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.500 to 1.206] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 2: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.6748, Regression, Cox; Hazard Ratio (HR) = 1.094, 95% CI 2-sided [0.720 to 1.662] — Hazard ratio for tirasemtiv vs placebo
Statistical Analysis 3: Comparison: Double-blind, Placebo-controlled: Group 1 - Placebo vs Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv; Test type: Superiority; p = 0.7694, Regression, Cox; Hazard Ratio (HR) = 0.938, 95% CI 2-sided [0.609 to 1.443] — Hazard ratio for tirasemtiv vs placebo

ADVERSE EVENTS:
Time Frame: AEs were collected from the first dose of open-label study drug through 28 days after the last dose of study drug.
Description: An AE was treatment-emergent if it started or worsened in severity after the first dose of study drug (in either the open-label [OL] or double-blind [DB] phases). The onset date of a TEAE in the OL phase that continued uninterrupted for ≥96 hours in the DB placebo-controlled phase was the date of the first dose of DB study drug.
  For patients randomized in the DB withdrawal phase, the onset date was on or before the last dose of study drug in the DB placebo-controlled phase.
Arm/Group | Open-label Lead-in: 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 1 - Placebo | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv | Double-blind, Withdrawal: Placebo | Double-blind, Withdrawal: Tirasemtiv to Placebo | Double-blind, Withdrawal: Tirasemtiv
All-Cause Mortality (participants affected / at risk) | 1/744 | 17/188 | 8/126 | 10/126 | 8/125 | 5/132 | 4/103 | 5/101
Serious Adverse Events (participants affected / at risk) | 11/744 | 53/188 | 30/126 | 30/126 | 32/125 | 15/132 | 15/103 | 11/101
Other Adverse Events (participants affected / at risk) | 640/744 | 182/188 | 125/126 | 125/126 | 125/125 | 123/132 | 100/103 | 95/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Lead-in: 250 mg Tirasemtiv (N=744) | Double-blind, Placebo-controlled: Group 1 - Placebo (N=188) | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv (N=126) | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv (N=126) | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv (N=125) | Double-blind, Withdrawal: Placebo (N=132) | Double-blind, Withdrawal: Tirasemtiv to Placebo (N=103) | Double-blind, Withdrawal: Tirasemtiv (N=101)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 9 | 12 | 7 | 2 | 2 | 4 | 3
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Euthanasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 4 | 0 | 2 | 2 | 0 | 3 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 4 | 2 | 0 | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 5 | 4 | 1 | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 4 | 2 | 1 | 3 | 3 | 3 | 0
Basal ganglia stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 3 | 1 | 0 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 5 | 6 | 6 | 3 | 3 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Lead-in: 250 mg Tirasemtiv (N=744) | Double-blind, Placebo-controlled: Group 1 - Placebo (N=188) | Double-blind, Placebo-controlled: Group 2 - 250 mg Tirasemtiv (N=126) | Double-blind, Placebo-controlled: Group 3 - 375 mg Tirasemtiv (N=126) | Double-blind, Placebo-controlled: Group 4 - 500 mg Tirasemtiv (N=125) | Double-blind, Withdrawal: Placebo (N=132) | Double-blind, Withdrawal: Tirasemtiv to Placebo (N=103) | Double-blind, Withdrawal: Tirasemtiv (N=101)
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 4 | 5 | 3 | 2 | 1 | 5
Constipation (Gastrointestinal disorders) | 21 | 40 | 24 | 21 | 27 | 17 | 15 | 13
Diarrhoea (Gastrointestinal disorders) | 24 | 19 | 7 | 10 | 9 | 5 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 10 | 14 | 8 | 8 | 7 | 7 | 5 | 8
Dysphagia (Gastrointestinal disorders) | 9 | 33 | 28 | 22 | 16 | 22 | 17 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 8 | 6 | 7 | 6 | 3 | 4 | 6
Nausea (Gastrointestinal disorders) | 108 | 30 | 20 | 38 | 26 | 9 | 7 | 6
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 19 | 14 | 9 | 3 | 14 | 5 | 11
Asthenia (General disorders) | 42 | 22 | 12 | 22 | 22 | 12 | 10 | 9
Fatigue (General disorders) | 204 | 61 | 43 | 54 | 50 | 32 | 32 | 23
Gait disturbance (General disorders) | 19 | 13 | 12 | 10 | 9 | 12 | 7 | 11
Oedema peripheral (General disorders) | 8 | 19 | 9 | 7 | 10 | 10 | 10 | 7
Peripheral swelling (General disorders) | 2 | 9 | 9 | 0 | 3 | 4 | 6 | 0
Nasopharyngitis (Infections and infestations) | 13 | 30 | 19 | 20 | 12 | 7 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 17 | 3 | 4 | 9 | 4 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 8 | 12 | 12 | 9 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 18 | 34 | 15 | 23 | 18 | 5 | 6 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 13 | 8 | 13 | 12 | 5 | 3 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 12 | 6 | 3 | 2 | 2 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 8 | 26 | 16 | 14 | 8 | 6 | 3 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 7 | 24 | 22 | 7 | 12 | 8 | 4 | 5
Traumatic fracture (Injury, poisoning and procedural complications) | 3 | 12 | 6 | 5 | 2 | 4 | 2 | 3
Weight decreased (Investigations) | 7 | 40 | 41 | 41 | 28 | 26 | 31 | 35
Decreased appetite (Metabolism and nutrition disorders) | 45 | 19 | 16 | 19 | 21 | 10 | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 14 | 4 | 7 | 4 | 8 | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 15 | 11 | 9 | 9 | 8 | 7 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 33 | 34 | 17 | 24 | 17 | 22 | 18 | 17
Muscular weakness (Musculoskeletal and connective tissue disorders) | 54 | 58 | 52 | 42 | 34 | 48 | 45 | 42
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 22 | 9 | 8 | 6 | 10 | 10 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 12 | 6 | 3 | 5 | 6 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 10 | 3 | 4 | 4 | 7 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 17 | 9 | 12 | 11 | 11 | 7 | 8
Balance disorder (Nervous system disorders) | 19 | 4 | 3 | 3 | 6 | 2 | 6 | 4
Dizziness (Nervous system disorders) | 361 | 45 | 47 | 55 | 56 | 11 | 21 | 15
Dysarthria (Nervous system disorders) | 30 | 18 | 15 | 8 | 12 | 13 | 11 | 10
Headache (Nervous system disorders) | 36 | 28 | 13 | 21 | 19 | 3 | 12 | 7
Muscle contractions involuntary (Nervous system disorders) | 11 | 9 | 15 | 8 | 12 | 5 | 5 | 7
Muscle spasticity (Nervous system disorders) | 11 | 4 | 5 | 10 | 6 | 4 | 7 | 7
Somnolence (Nervous system disorders) | 90 | 14 | 19 | 19 | 18 | 3 | 5 | 10
Tremor (Nervous system disorders) | 22 | 4 | 4 | 13 | 11 | 5 | 5 | 3
Affect lability (Psychiatric disorders) | 8 | 6 | 5 | 5 | 6 | 8 | 2 | 5
Anxiety (Psychiatric disorders) | 15 | 19 | 14 | 13 | 24 | 13 | 15 | 10
Depression (Psychiatric disorders) | 21 | 22 | 8 | 24 | 23 | 14 | 9 | 14
Insomnia (Psychiatric disorders) | 31 | 25 | 23 | 25 | 30 | 19 | 19 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 26 | 12 | 16 | 7 | 12 | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 35 | 17 | 22 | 18 | 22 | 13 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 12 | 11 | 7 | 8 | 5 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 6 | 6 | 7 | 6 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 8 | 9 | 12 | 3 | 8 | 3 | 5 | 3
Parathesia (Nervous system disorders) | 6 | 3 | 4 | 1 | 8 | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 9 | 6 | 6 | 3 | 7 | 3 | 4 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 5 | 8 | 2 | 4 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 2 | 2 | 7 | 2 | 3 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 10 | 5 | 4 | 3 | 7 | 3 | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 6 | 3 | 3 | 4 | 4 | 6 | 0
Vertigo (Ear and labyrinth disorders) | 19 | 7 | 13 | 7 | 4 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02496767/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02496767/SAP_001.pdf